CLINICAL TRIAL: NCT00198692
Title: Randomized Clinical Trial of Self-Management Educational Program for Persons With Limb Loss.
Brief Title: Self-Management Program for Persons With Limb Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: University of Washington (Other); Amputee Coalition of America (Other)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: R04/CCU322981-02
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-10-28 (Estimated); Status verified 2005-09

CONDITIONS: Amputation; Depression; Pain; Anxiety
Keywords: amputation; depression; pain; anxiety; self-management; secondary conditions
MeSH Terms: conditions — Depression; Pain; Anxiety Disorders | interventions — Self-Management

INTERVENTIONS:
Behavioral: self-management

SUMMARY:
The specific aims of this study are:

1. To develop and pilot a self-management (SM) intervention for persons with limb loss in a group setting using a participatory action research (PAR) strategy.
2. To evaluate the feasiablity and effectiveness of a SM intervention within the context of the existng network of limb loss peer support groups

   Hypothesis #2a: The SM intervention groups will be more effective than standard support group activities in reducing pain, depression and anxiety, and increasing positive mood and improving function and overall quality of life.

   Hypothesis #2b: Improvements in pain, depression, anxiety, function and quality of life will correlate strongly with improvements in self-efficacy, catastrophizing, and satisfaction with the prosthesis and prosthetic services.

   Hypothesis #2c: Gains in outcome will be maintained for one year.

   Hypothesis #2d: Characteristics of study participants and their environment (i.e. sociodemographics, co-morbidities, economic and educational resources, hope, and social support) will correlate with outcome and mediate the effect of the intervention.
3. To determine the costs of the intervention and examine the relationship between costs and effectiveness.

Hypothesis #3a: When compared to the control support group, the SM intervention will be cost-effective in terms of gains in quality adjusted years of life.

DETAILED DESCRIPTION:
Approximately 1.2 million Americans are living with limb loss. Pain, psychological distress, reduced function and disability are common conditions following limb loss and are related to reduced quality of life. Our own work has identified depression, anxiety, and pain as significant problems for community dwelling persons with limb loss. Traditionally, interventions for disabling impairments and related secondary conditions focus on standard medical treatments such as medication, surgery or rehabilitative therapies. Self-management (SM) interventions, on the other hand, have been found to be effective in reducing secondary conditions and disability associated with some chronic conditions using individual and group-based delivery methods. To date, no SM intervention has been developed for, and evaluated in, persons with limb loss. The goal of the project is to develop and test the efficacy of a community-based self-management intervention for reducing pain, depression, and anxiety and improving positive mood, self-efficacy and function in persons with limb loss. The intervention will build on the already exisitng national network of community-based peer support groups developed by the Amputee Coalition of America (ACA). Establishing the efficacy of commmunity-based SM interventions for persons with limb loss has the potential to improve the health and quality of life for this population

ELIGIBILITY:
Inclusion Criteria:

* Persons with acquired or congenital limb loss

Exclusion Criteria:

* Non-English speakers

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2003-08; Study Completion 2006-03

PRIMARY OUTCOMES:
The primary outcome measures are pain, anxiety, depression, and positive mood.

SECONDARY OUTCOMES:
Secondary outcome measures are restrictions in activities and participation and health related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Ellen J MacKenzie, PhD, Principal Investigator — Johns Hopkins University Bloomberg School of Public Health
Locations (1):
- Johns Hopkins University Bloomberg School of Public Health, Baltimore, Maryland, United States